CLINICAL TRIAL: NCT02478203
Title: Intubation on a Pediatric Manikin by Emergency Medical Staff: a Comparison of Direct Laryngoscopy, Airtraq and Glidescope in Normal, Tongue Edema and Face-to-face Intubation Models
Brief Title: Intubation on a Paediatric Manikin by Emergency Staff: a Comparison of Airtraq and Glidescope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2014/108
Record Dates: First submitted 2015-04-17; First posted 2015-06-23 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Difficult Intubation
Keywords: Airtraq; Glidescope; pediatric; face-to-face

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- normal (Placebo Comparator): intubation of a normal airway pediatric manikin with direct laryngoscopy, airtraq , glidescope
  Interventions: Device: Airtraq; Device: Glidescope; Device: direct laryngoscopy
- tongue edema (Active Comparator): intubation of a tongue edema simulated pediatric manikin with diract laryngoscopy, glidescope and airtraq
  Interventions: Device: Airtraq; Device: Glidescope; Device: direct laryngoscopy
- face-to-face intubation (Active Comparator): intubation of an entrapped pediatric manikin with diract laryngoscopy, glidescope and airtraq
  Interventions: Device: Airtraq; Device: Glidescope

INTERVENTIONS:
Device: Airtraq — videolaryngoscope for difficult airway
Device: Glidescope — videolaryngoscope for difficult airway
Device: direct laryngoscopy — gold standart for intubation
  Arms: normal; tongue edema

SUMMARY:
After Local Human Research Ethics Committee approval, emergency medical staff enrolled in this study. After watching a video about the intubation using Airtraq, Glidescope or direct laryngoscopy, they attempted to intubate a pediatric manikin in three different airway models.

DETAILED DESCRIPTION:
After Local Human Research Ethics Committee approval, emergency medical staff enrolled in this study. After watching a video about the intubation using Airtraq , Glidescope or direct laryngoscopy, they attempted to intubate a pediatric manikin in three different airway models; normal airway, tongue edema and an entrapped model by face-to-face approach. Intubation attempts, insertion and intubation times, success rates, Cormack-Lehane grades and the need for maneuvers of these devices were recorded.

ELIGIBILITY:
Inclusion Criteria:

* pediatric

Exclusion Criteria:

* adult

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
intubation time | 120 seconds
  handling of the device till visualization of the tube entering through the vocal cords

SECONDARY OUTCOMES:
need of maneuvers (mender applied or not) | intraoperative
  maneuver applied or not
esophageal intubation (eosophageal intubation occured or not) | intraoperative
  eosophageal intubation occured or not
intubation attempts (is it increased or not) | intraoperative
  the patient intubated at which attempt?
cormack-lehane grade (which one improves the cormack- lehane grade) | intraoperative
insertion time | 30 seconds
  handling of the device till the glottic visualization

CONTACTS AND LOCATIONS:
Overall Officials: Zehra I Arslan, Study Director — Anesthesiology and Reanimation
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)